CLINICAL TRIAL: NCT03780920
Title: Interest of an Early Osteopathic Treatment in Infants in the Prevention of Cranial Deformations : Positional Plagiocephaly and Brachycephaly.
Brief Title: Preventive Osteopathic Treatment of Plagiocephaly
Acronym: TOPP PLAGIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RECHMPL18_0207
Record Dates: First submitted 2018-12-13; First posted 2018-12-19 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Positilonal Deformation of the Skull; Head Turn Preference; Axial Hypertony
MeSH Terms: interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osteopathic treatment (Active Comparator)
  Interventions: Procedure: manual therapy/osteopathy
- Control group (No Intervention)

INTERVENTIONS:
Procedure: manual therapy/osteopathy — In this group, children will benefit from early osteopathic treatment over a period ranging from the third day to 4 months. The number of sessions will not be fixed, on average, 3 sessions will be carried out during this period at the University Hospital of Montpellier.
  The duration of the session will be between 20 minutes to 30 or even 40 minutes
  Arms: Osteopathic treatment

SUMMARY:
Positional cranial deformities (PCD), plagiocephaly and brachycephaly are a common reason for pediatric consultation, which has increased significantly since the recommendation to lay babies on their backs to prevent unexpected infant death (ILD). CPD is a source of concern for parents about their impact on psychomotor development and the aesthetic risk of deformity. The High Authority for Health (HAS) will soon put in place recommendations with a fact sheet for health professionals and the public. The aim of this research is to study whether early treatment of rotation disorders and hypertonia in newborns by manual osteopathic techniques would prevent the occurrence of positional deformities of the skull.

The main objective is to evaluate the effectiveness of an early osteopathic treatment on the rate of CPP (plagiocephalic and postural brachycephalia) at 4 months in newborns at risk.

the secondary objective is: to evaluate the effectiveness of an early osteopathic treatment on the quality of life of the child at 4 months.

Methodology: Controlled, randomized monocentric two-arm parallel study between (1) osteopathic follow-up and (2) osteopathy-free follow-up. The inclusion period will be 18 months and the follow-up period is 4 months.

Procedure: The two groups will be evaluated at 3 days and 4 months. The experimental group will benefit from an osteopathic treatment of 3 days of life to 4 months with a frequency of 3 to 4 sessions. Both groups will benefit from sleeping, carrying, positioning and stimulation advice.

The perspectives are:

* the decrease in the prevalence of CPP after early osteopathic treatment.
* Defining a decision algorithm for early osteopathic treatment.
* Subject to recommendations on the indication of early osteopathic treatment in neonates at risk.

ELIGIBILITY:
Inclusion Criteria:

* Newborn baby aged 3 days and until the maternity leave
* Newborn with at least one risk factor for cranial deformity:

  * Newborn who received instrumental vaginal delivery.
  * Newborn presenting:

    * a preferential side,
    * global axial hypertonia,
    * Localized suboccipital hypertonia
  * Newborn presenting:

    * cranial deformity at birth,
    * a deformation of the face,
    * deformity of the trunk in scoliosis, comma or hyperextension

Exclusion Criteria:

* Newborn with congenital muscular torticollis (managed directly in physiotherapy)

  * Premature neonate (<37SA)
  * Newborn with a malformation pathology
  * Newborn with craniosynostosis.
  * Newborn with a contraindication to the practice of osteopathy.

Ages: 3 Days to 11 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
Positionnal skull deformation : plagiocephaly and brachycephaly | four month
  cranial vault asymetry index and cranial index measured with caliper between the age of 3 to 10 days and at 4 months measured blind of the randomization arm

SECONDARY OUTCOMES:
Questionnaire QUALIN | fourth month
  the"questionnaire QUALIN" is a quality of life assessment questinniare for infant under 3 months of age, valided in Europe(French, Spanish, English and Italian)

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume CAPTIER, Pr, Principal Investigator — University Hospital, Montpellier
Locations (1):
- CHU Arnaud de Villeneuve, Montpellier, Hérault, France